CLINICAL TRIAL: NCT01483937
Title: Clinical Trial Evaluation of a Sensory Enrichment Multimodal Device (SEMD) on Physical Therapy Patients With Disequilibrium
Brief Title: Evaluation of a Sensory Enrichment Multimodal Device (SEMD) on Physical Therapy Patients With Disequilibrium
Acronym: SEMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karen L Atkins (Industry)
Responsible Party: Sponsor-Investigator, Karen L Atkins, Study Director, BalanceSense LLC
Organization: BalanceSense LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10-221:1.2; W81XWH-10-C-0184-01 (Other Grant/Funding Number: OSD-Army)
Record Dates: First submitted 2011-11-30; First posted 2011-12-02 (Estimated); Results first posted 2014-06-27 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-06

CONDITIONS: Vestibular Diseases; Labyrinth Diseases; Ear Diseases; Otorhinolaryngologic Diseases; Traumatic Brain Injury
Keywords: Keywords provided by BalanceSense, LLC:; Physical Therapy; Rehabilitation; Disequilibrium; Balance dysfunction or disorder; Vestibular; Mild Traumatic Brain Injury (mTBI); Vibrotactile
MeSH Terms: conditions — Vestibular Diseases; Labyrinth Diseases; Ear Diseases; Otorhinolaryngologic Diseases; Brain Injuries, Traumatic; Dysequilibrium syndrome; Brain Concussion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care physical therapy only (Active Comparator): Subjects will receive usual care physical therapy intervention provided by vestibular and balance specialists. Usual care physical therapy, in general, includes but is not limited to static and dynamic balance activities with or without head movements on firm floor or compliant surfaces.
  Interventions: Other: Usual care physical therapy only
- Usual care physical therapy plus SEMD (Experimental): Subjects will receive usual care physical therapy intervention provided by vestibular balance specialists while using the Sensory Enrichment Multimodal Device (SEMD). SEMD protocols use visual, vibrotactile, and auditory cueing referenced to subject's Center of Gravity (COG) and/or Sum of Pressure (SOP) data collected from a force platform upon which the subject is placed. Static and dynamic balance activities with or without head movement are preformed while watching a computer screen; paced with an auditory metronome; and cued by "touch" vibration via coin tactors imbedded in a belt worn around the waist matching the COG/SOP data display.
  Interventions: Device: Usual care physical therapy plus SEMD

INTERVENTIONS:
Device: Usual care physical therapy plus SEMD — Patients will receive usual care physical therapy while wearing SEMD. SEMD protocols will also be provided to device subjects.
  Other Names: BalanceSense
  Arms: Usual care physical therapy plus SEMD
Other: Usual care physical therapy only — Subjects will receive usual care physical therapy from vestibular and balance specialists.
  Arms: Usual care physical therapy only

SUMMARY:
Purpose of this study is to determine the efficiency and safety of a Sensory Enrichment Multimodal Device (SEMD) when applied in conjunction with usual care vestibular-balance physical therapy for rehabilitation of patients who fall as a result of vestibular inducted disequilibrium.

Study participants will receive regular physical therapy, and some will use the SEMD device while receiving usual care vestibular-balance physical therapy. The device is an elastic belt that holds eight small battery powered vibrating disks. When using the device, you will sit or stand on a force platform that measures body sway. That movement information is sent to a computer which then sends the information to you via the vibrating disks. The vibrating disks are similar to a vibrating cell phone: you can feel the vibration but it is not uncomfortable. You can also see your sway movement on the computer screen. Some tests and activities will be paced with a beeping sound.

The aim of this study is six-fold: 1. Demonstrate the relative efficiency between SEMD and conventional vestibular-balance physical therapy as reported by treating physical therapists' by counting number of skills acquired in a treatment session, and the amount of time needed to acquire the skill; 2. Demonstrate greater improvement earlier on in balance test scores when using the SEMD as an adjunct to conventional vestibular-balance physical therapy; 3. Determine the difference in vestibular habituation between physical therapy plus SEMD and conventional vestibular-balance physical therapy; 4. Demonstrate a more immediate reduction in fall occurrence when using SEMD as an adjunct to conventional vestibular-balance physical therapy; 5. Determine the patient's perception of quality of life between physical therapy plus SEMD and conventional vestibular-balance physical therapy; 6. Determine difference in acquisition of large movement tasks of tandem walk, step quick-turn, and kneel-shoulder rifle-return to stand between subjects that have trained with SEMD and conventional vestibular-balance physical therapy .

In addition to primary and secondary outcome measurements, efficiency of skill acquisition, devised for this study, will be evaluated by tracking the number of skills and length of time needed to acquire each skill for each physical therapy session using the Patient Skill Acquisition Chart (PSAC). Usefulness of Tandem Walk, Step Quick-turn, and Kneel- Shoulder Rifle-Return to Stand as intervention outcome, also devised for this study, will be evaluated with pre test to post tests Modified Functional Independence Measure - Motor (MFIM-Motor). These measurements were devised for this study, and will be evaluated for informational purposes only.

DETAILED DESCRIPTION:
This study will compare two approaches of physical therapy intervention within vestibular deficit populations that frequently fall: 1. physical therapy plus SEMD, and 2. usual care physical therapy only.

Multimodal sensory cueing gives additional or enriched information to complement postural and mobility decisions. SEMD displays combine vibrotactile, visual and audio cueing that are intuitive and non-intrusive within a balance training system.

Study intervention includes a maximum of 12 physical therapy intervention sessions, 2 times per week for 6 weeks or normalization of SOT, whichever occurs first. Usual care physical therapy prescriptions are written specific for number of sessions over a specific duration of time. Discharge from physical therapy occurs when number of sessions within a specified period of time is exhausted or goals specified by the physical therapist are met. Data collection includes 1 pre test and 4 post tests at intervals during the weeks of intervention, plus 3 follow-up phone interviews at specified intervals after intervention for maximal study duration of 6 months. A patient must attend at least 4 physical therapy intervention sessions for their data to be used and for the follow-up phone interviews to be initiated.

ELIGIBILITY:
Inclusion Criteria:

1. Self-reporting 2 or more falls with or without injury within the past 6 months.
2. Below normal SOT containing a abnormal vestibular score.
3. Potential to benefit from physical therapy as indicated by physician prescription referral.
4. Able to sit and to stand unaided for 2 minutes.
5. Willing and able to complete all testing, training, and follow-up evaluations required by the study protocol.

Exclusion Criteria:

1. Fluctuating Meniere's
2. Vestibular injury requiring surgery such as perilymph fistula
3. Moderate progressive neurologic disease such as multiple sclerosis
4. Does not speak and understand the English language
5. Resides in a nursing home
6. Unable to provide own consent.

Ages: 21 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-11; Primary Completion 2013-05 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen L Atkins, PhD, PT, Study Director — BalanceSense LLC
Locations (4):
- United States (4):
  - England Physical Therapy, Garden Grove, California
  - Florida Ear & Balance Center, Celebration, Florida
  - Stevenson & Associates Physical Therapy, Fort Myers, Florida
  - Brooks Balance Center, Jacksonville, Florida

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment continued for one year resulting in 39 subjects pre screened for inclusion in the study.
Pre-assignment Details: Seven subjects who had signed Informed Consent prior to inclusion/exclusion screening failed screening: thirty-two subjects participated in the physical therapy protocol.
Groups:
- Conventional Care Physical Therapy Only: Subjects received usual physical therapy intervention provided by vestibular and balance specialists.
- Conventional Physical Therapy Plus SEMD: Subjects received usual physical therapy intervention while using SEMD: SEMD protocols augmented conventional physical therapy.
Period: Overall Study
Arm/Group | Conventional Care Physical Therapy Only | Conventional Physical Therapy Plus SEMD
Started | 15 | 17
Completed | 11 | 14
Not Completed | 4 | 3
Not completed — Withdrawal by Subject | 4 | 3

BASELINE CHARACTERISTICS:
Population: 4 withdrew from Conventional care physical therapy 3 withdrew from Conventional care physical therapy plus SEMD
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional Care Physical Therapy Only | Conventional Physical Therapy Plus SEMD | Total
Number analyzed (Participants) | 11 | 14 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 1 | 4
  >=65 years | 8 | 13 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.44 (10.00) | 73.35 (7.46) | 71.64 (8.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 17
  Male | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 11 | 14 | 25

OUTCOME MEASURES:

1. Primary Outcome: Assessment of the Efficacy of the SEMD Device in Improving Vestibular Function Was Evaluated With Change in Pre Test to Post Test 1 Sensory Organization Test (SOT).
Description: Sensory Organization Test (SOT) is a standing balance test that measures the subject's ability to control postural sway under vestibular, visual, and somatosensory conflict. Score ranges from 0 to 100 with higher score indicating better control of postural sway.
Time Frame: Pre Test to Post Test 1 after two physical therapy sessions (one week)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Conventional Care Physical Therapy Only | Conventional Physical Therapy Plus SEMD
Number analyzed (Participants) | 11 | 14
units on a scale | 9.82 (10.68) [-17.5 to -1.1] | 7.29 (9.33) [-25.7 to -7.1]
Statistical Analysis 1: Comparison: Conventional Care Physical Therapy Only vs Conventional Physical Therapy Plus SEMD; Test type: Superiority or Other; p = .533, ANOVA

2. Primary Outcome: Assessment of the Efficacy of the SEMD Device in Improving Vestibular Function Was Evaluated With Change in Post Test 1 to Post Test 2 Sensory Organization Test (SOT).
Description: as for outcome 1
Time Frame: Post Test 1 to Post Test 2 after four physical therapy sessions (two weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Conventional Care Physical Therapy Only | Conventional Physical Therapy Plus SEMD
Number analyzed (Participants) | 11 | 14
units on a scale | 9.36 (12.80) | 5.00 (8.49)

3. Primary Outcome: Assessment of the Efficacy of the SEMD Device in Improving Vestibular Function Was Evaluated With Change in Post Test 2 to Post Test 3 Sensory Organization Test (SOT).
Description: as for outcome 1
Time Frame: Post Test 2 to Post Test 3 after eight physical therapy sessions (4 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Conventional Care Physical Therapy Only | Conventional Physical Therapy Plus SEMD
Number analyzed (Participants) | 11 | 14
units on a scale | 3.27 (7.94) | 8.86 (7.72)

4. Primary Outcome: Assessment of the Efficacy of the SEMD Device in Improving Vestibular Function Was Evaluated With Change From Post Test 3 to Post Test 4 Sensory Organization Test (SOT).
Description: as for outcome 1
Time Frame: Post Test 3 to Post Test 4 after twelve physical therapy sessions (6 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Conventional Care Physical Therapy Only | Conventional Physical Therapy Plus SEMD
Number analyzed (Participants) | 11 | 14
units on a scale | 5.09 (6.70) | .86 (6.57)

5. Secondary Outcome: Percent of Subjects Decreasing Fall Risk Measured by Functional Gait Assessment Pre Test to Post Test 2
Description: Functional Gait Assessment is a 10-item gait assessment based on the Dynamic Gait Index. Requirements: A marked 20 foot walkway that is marked with a 12 inch width. Scoring: a four-point ordinal scale, ranging from 0-3 where "0" indicates the lowest level of function and "3" the highest level of function. Total Score = 30 with higher score indicating safer ambulation with lower risk of falling.
  Criterion Validity: "Authors support a cut off score of 23/30 for independent safe ambulation".
  Interpretation: 1) 0-19 is predictive of falls in the elderly. 2) 20-22 indicates likelihood of unexplained fall in community-dwelling, older adults, and predictive of likelihood of falling in patients with vestibular disorders.
  3) 23-30 = safe ambulators
Time Frame: Pre Test to Post Test 2 after four physical therapy sessions within 10 days
Measure: Number; unit: percentage of participants
Arm/Group | Conventional Care Physical Therapy Only | Conventional Physical Therapy Plus SEMD
Number analyzed (Participants) | 11 | 14
percentage of participants | 20 (2.38) | 77 (2.01)

6. Secondary Outcome: Percent of Subjects Reporting Decrease in Self-report Fall(s) Occurrence Pre Test to Post Test 1
Description: A fall is an unintentional change in position causing an individual to land at a lower level, on an object, the floor, the ground or other surface with or without injury. This includes: slips, trips, falling into other people, being lowered, loss of balance, and legs giving way. (Exclude sudden onset of paralysis, epileptic seizure, or overwhelming external force.)
Time Frame: Pre Test to Post Test 1 after 2 physical therapy sessions within 4 days
Measure: Number; unit: percentage of participants
Groups:
- Conventional Care Physical Therapy Only: Subjects received usual physical therapy intervention provided by vestibular and balance specialists.
  Conventional physical therapy only: Subjects received standard care physical therapy from vestibular and balance specialists.
- Conventional Physical Therapy Plus SEMD: Subjects received usual physical therapy intervention while using SEMD: SEMD protocols augmented conventional physical therapy.
  Usual care physical therapy plus SEMD: Patients received standard care physical therapy while wearing SEMD. SEMD protocols were provided to device subjects.
Arm/Group | Conventional Care Physical Therapy Only | Conventional Physical Therapy Plus SEMD
Number analyzed (Participants) | 11 | 14
percentage of participants | 9 | 54

7. Secondary Outcome: Percent of Subjects Decreasing Fall Risk Measured by Berg Balance Scale Pre Test to Post Test 2
Description: Berg Balance Scale Description: 14-item scale designed to measure balance of the older adult in a clinical setting, and measures mobility related to activities of daily living. Description: This 14-item performance-based instrument is intended for individuals with some degree of balance impairment.
  Scoring: A five-point ordinal scale, ranging from 0-4. "0" indicates the lowest level of function and "4" the highest level of function. Total Score = 56 with higher score indicting safer ambulation with lower risk of falling.
  Criterion Validity: "Authors support a cut off score of 45/56 for independent safe ambulation".
  Interpretation: 41-56 = low fall risk 21-40 = medium fall risk 0 -20 = high fall risk
  Riddle and Stratford, 1999, examined 45/56 cutoff validity and concluded:
  * Sensitivity = 64% (Correctly predicts fallers)
  * Specificity = 90% (Correctly predicts non-fallers)
Time Frame: Pre Test, Post Test 2 after 4 physical therapy sessions within 10 days.
Measure: Number; unit: percentage of participants
Groups:
- Conventional Care Physical Therapy Only: Subjects received usual physical therapy intervention provided by vestibular and balance specialists.
  Conventional physical therapy only: Subjects received usual care physical therapy from vestibular and balance specialists.
Arm/Group | Conventional Care Physical Therapy Only | Conventional Physical Therapy Plus SEMD
Number analyzed (Participants) | 11 | 14
percentage of participants | 43 | 100

8. Secondary Outcome: Self-rated Disability Measured by Vestibular Rehabilitation Benefit Questionnaire Pre Test to Post Test 4
Description: Vestibular Rehabilitation Benefit Questionnaire asks the patient to self-rate disability as it affects their quality of life. Scale goes from zero, no disability, to 100 or maximal disability. The Total Benefit includes two subsets: 1) dizziness symptoms, and 2) quality of life.
Time Frame: Pre test to Post Test 4 or 12 Physical Therapy sessions within 42 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Conventional Care Physical Therapy Only | Conventional Physical Therapy Plus SEMD
Number analyzed (Participants) | 11 | 14
units on a scale
  Pre Test | 39.14 (17.95) | 34.30 (6.52)
  Post Test 4 | 31.27 (8.25) | 28.32 (11.10)

9. Secondary Outcome: Head Shake Sensory Organization Test (HS_SOT)
Description: Head Shake Sensory Organization Test (HS-SOT)
  HS-SOT instructs the patient to static stand shoulder width apart with eyes closed and uses the SOT Condition 5 sway surface protocol while shaking the head horizontally 120 degrees per second. This protocol is safe for patients when they have normalized all SOT scores. Because study subjects were reaching SOT normalization after Post Test 2, the data collected was scant and not suitable for analysis.
Time Frame: Pre Test, Post Test 1 and Post Test 4
Arm/Group | Conventional Care Physical Therapy Only | Conventional Physical Therapy Plus SEMD
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Conventional Care Physical Therapy Only | Conventional Physical Therapy Plus SEMD
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/17
Other Adverse Events (participants affected / at risk) | 0/15 | 0/17

LIMITATIONS AND CAVEATS:
Small number of subjects recruited because of lengthy study commitment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No